CLINICAL TRIAL: NCT06318195
Title: Internet Delivered Condensed Cognitive Behavioral Treatment (Prolonged Exposure) for Individuals Treated Within Somatic Trauma Care.
Brief Title: Condensed Digital Prolonged Exposure for Individuals Treated Within Somatic Trauma Care.
Acronym: CiPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Maria Bragesjo, PhD, Licensed Psychologist, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-06821-01
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Post Traumatic Stress Disorder; Acute Stress Disorder
Keywords: condensed prolonged exposure; Internet-delivered; PTSD; trauma; early intervention; prevention; CIPE
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Prolonged exposure will be offered in a brief digital format with therapist support for three weeks. Treatment comprises of psychoeducation, rationales, in vivo exposure, imaginal exposure and relapse prevention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Condensed Internet delivered prolonged exposure (CIPE) (Experimental): Condensed Internet delivered prolonged exposure (CIPE) for three weeks with therapist support.
  Interventions: Behavioral: Condensed Internet delivered prolonged exposure (CIPE)

INTERVENTIONS:
Behavioral: Condensed Internet delivered prolonged exposure (CIPE) — Condensed Internet delivered prolonged exposure (CIPE) with therapist support for three weeks.

SUMMARY:
The purpose of the study is to investigate the feasibility of implementation aspects, treatment effects and change processes regarding a brief trauma-focused Internet-based CBT treatment, for patients who have been treated in trauma care at Karolinska University Hospital and who exhibit symptoms of psychological consequences of the traumatic event. Another aim is to explore factors (predictors, moderators and mediators) that influence the effect of the treatment, in order to better understand who responds to the treatment.

DETAILED DESCRIPTION:
The study is un-controlled with 250 participants that will undergo a brief trauma-focused Internet-based CBT treatment, delivered as a three-week treatment comprising of four modules (psychoeducation/rational, in vivo exposure, imaginal exposure and relapse prevention). The primary outcome is the PCL-5. Secondary outcomes are level of depression (PHQ-9), quality of life (WSAS) and predictors, moderators and mediators of clinically meaningful change in symptoms, dropout rate, rates of inclusion, attrition, adherence,and negative effects.

Self-reported, qualitative data from participants will be gathered at treatment completion to capture participants' experiences of participating in the intervention, as well as their views on how to further improve the intervention. The treatment effects will be evaluated using a within-group design with repeated measurements. Participants in the study will be will recruited from patients treated in the somatic trauma care at the Karolinska University Hospital in Stockholm, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to trauma in the past two months according to criterion A for PTSD in the DSM-5 (exposed to death, threatened death, actual or threatened serious injury, or actual or threatened sexual violence).
* PCL-5 total sum score>10
* ≥ 18 years
* Situated in Sweden
* Signed informed consent

Exclusion Criteria:

* Other serious comorbidity as primary concern (ongoing substance dependence, untreated bipolar disorder, psychotic symptoms, severe depression, borderline personality disorder, high suicidal risk according to the MINI)
* Unable to read and write in Swedish
* Receiving other psychological trauma-focused treatment
* Ongoing trauma-related threat (e.g., living with a violent spouse)
* Not stable dose of antidepressant medication the last two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms as assessed by the PTSD Check List - DSM-5 (PCL-5) | week -3, -2 and -1 before treatment start, immediately before start of treatment, weekly through three weeks of treatment, post-treatment (immediately after treatment completion at three weeks), and the 1 month and 6 months follow up.
  The PCL-5 is a 20-item self-report measure based upon the Diagnostic and Statistical Manual (DSM-5) criteria for PTSD. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.

SECONDARY OUTCOMES:
Change in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) | week -3 before treatment start, immediately before start of treatment, weekly through three weeks of treatment, post-treatment (immediately after treatment completion at three weeks), and the 1 month and 6 months follow up.
  The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms. Scores are calculated based on how frequently a person experiences 9 symptoms of depression ranging from "not at all" response is scored as 0; "several days" response is 1; "more than half the days" response is 2; and "nearly every day" response is 3. Higher scores represents more depressive symptoms.
Change in psychosocial impairment measured by The Work and Social Adjustment Scale (WSAS), adapted to symptoms of post-traumatic stress. | week -3 before treatment start, immediately before start of treatment, , weekly through three weeks of treatment, post-treatment (immediately after treatment completion at three weeks), and the 1 month and 6 months follow up.
  WSAS is a short, self-reported instrument consisting of five items about psychosocial impairments rated on a nine-point Likert scale. A higher score means more severe impairment.

OTHER OUTCOMES:
Participants satisfaction with treatment. | Immediately after treatment completion.
  Qualitative questions pertaining participants satisfaction with the treatment.
Adverse events related to treatment. | Immediately after treatment completion.
  Adverse events related to treatment measured by with a free text option where participant is instructed to describe the possible event in detail. If the participant reported any adverse event, additional follow-up questions about intensity, duration etc. will also be given.
Number of completed treatment modules | Baseline up to 3 weeks
  Data will be gathered on total number of completed modules during the three week treatment.
Number of messages sent and received in the digital platform | Baseline up to 3 weeks
  Data will be gathered on total number of messages sent and received in the digital platform during the three week treatment.
Number of completed home work assignments by the participant during the treatment period | Baseline up to 3 weeks
  Data will be gathered on total number of completed home work assignments by the participant during the three week treatment.
The proportion of participants that conducts the weekly measures and further assessment points | Baseline up to 6 months
  The proportion of participants that conducts the weekly measures and further assessment points
The proportion of participants that go through the entire treatment period | Baseline up to three weeks
  The proportion of participants that go through the entire treatment period
Number of drop-outs from treatment | Baseline up to three weeks
  Number of drop-outs from treatment
Rates of inclusion to the study | Baseline
  Data on rates of inclusion will be considered as an indication of the feasibility of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bragesjö, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Universitetssjukhuset; Tema Kvinnohälsa och Hälsoprofessioner; Medicinsk Enhet Medicinsk Psykologi; Sektion Beteendemedicin, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No